CLINICAL TRIAL: NCT05356975
Title: The Effects of Eight Weeks of Virtual Training Based on Supersets vs. Concurrent Training on Muscle Strength, Cardiorespiratory Fitness, Motivation, Adherence, and HRQL in Women With Low to Moderate Levels of Physical Activity.
Brief Title: Virtual Training Based on Supersets vs. Concurrent Training in Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Victor Hugo Arboleda Serna, Principal Investigator, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Virtual Superset-UdeA
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers
Keywords: Resistance training; Superset resistance training; Concurrent training; Virtual training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superset (Experimental): This group will perform three strength circuit training. Each circuit training consists of three exercises (lower, middle, and upper body exercises) performed in a supersets fashion. This order makes it less complex, which is important given the characteristics of the population.
  Interventions: Behavioral: Superset
- Concurrent (Active Comparator): This group will perform six resistance exercises in a traditional fashion (three exercises for the lower body, three exercises for the upper body) and three aerobic exercises (floor tap squat, jumping jacks, and skaters).
  Interventions: Behavioral: Concurrent

INTERVENTIONS:
Behavioral: Superset — A strength circuit training will be performed in a supersets fashion. Three strength circuit training in three blocks.
  1. One leg squat, side plank, and push up.
  2. Deadlift, lumbar extension stretch, and row.
  3. Glute bridge, crunches, and front raise.
  Arms: Superset
Behavioral: Concurrent — Six resistance exercises in a traditional fashion: three exercises for the lower body (one leg squat, deadlift, and glute bridge). Three exercises for the upper body (push up, row, and front raise). And three aerobic exercises (floor tap squat, jumping jacks, and skaters).
  Arms: Concurrent

SUMMARY:
There are different forms of physical activity proven to improve muscular strength and cardiorespiratory fitness. One of them is concurrent training, which is defined as the combination of two or more physical capacities in the same session (resistance and endurance training). Another modality is superset training, which is characterized by performing two or more exercises for the same muscle group, or a different muscle group, consecutively, with minimal recovery between them.

To date, the evidence has shown studies comparing different resistance training protocols, vs. aerobic training, and vs. concurrent training, performed in various ways, on muscle strength and cardiorespiratory fitness. Most of these studies involved men with resistance training experience, and little research linked women. It should be noted that no study found has used virtual training to test the effects of superset training compared to concurrent training in women with low to moderate levels of physical activity.

Therefore, this study aims to identify the effect of a superset training program vs. a concurrent training program on muscle strength, cardiorespiratory fitness, motivation, adherence, and health-related quality of life in women with a low to moderate level of physical activity for eight weeks virtually.

DETAILED DESCRIPTION:
Sixty women will be randomly assigned to two groups (superset and concurrent). The interventions will be carried out virtually asynchronously, only sessions 1, 5, 9, 13, 17, and 21 will be supervised synchronously. Follow-up will be done through WhatsApp messages. Both groups will have a training frequency of 3 times a week for eight weeks. In the training sessions, strength exercises with self-loading (crunches, one leg squat, side plank, push up, deadlift, lumbar extension stretch, row, glute bridge, front raise) and/or aerobic exercises (floor tape squat, jumping jacks, skaters). Each group will execute the same number of series and repetitions during the 8 weeks, the performance of strength exercises will be standardized at 45 bpm throughout the protocol, and aerobic exercises at 70 bpm. Intensity will be controlled by resting between sets, starting with 90 seconds in week one, decreasing by 15 seconds every two weeks until reaching 45 seconds.

Each participant will have initial and final evaluations to measure muscle strength in lower, middle, and upper kinetic chains. Queen's College test will be used to assess cardiorespiratory fitness, BREQ-2, and SF-12 questionnaires will be used to measure motivation and health-related quality of life respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Physical activity (<600 to ≤1500 MET/min/wk)

Exclusion Criteria:

* Diabetes
* Hypertension
* History of cardiovascular disease
* History of coronary heart disease
* Osteoporosis
* Pregnancy
* Breast-feeding women
* Psychological, neuromotor, and/or osteo-muscular conditions that may affect participation in an exercise program.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in muscular strength | Baseline and 8-weeks
  Test: One leg squat, leg lever, and push up. A maximum number of repetitions as possible to failure.

SECONDARY OUTCOMES:
Cardiorespiratory fitness | Baseline and 8-weeks
  Queens College Step Test
  The test consists of 3 minutes of stepping up and down on a 41.3 cm step at a set rate of 22 steps per minute for females and at 24 steps per minute for males. Estimation of VO2max can be calculated from the test results as follow:
  Men: VO2max(ml/kg/min) = 111.33 - (0.42 x heart rate (bpm) Women: VO2max(ml/kg/min) = 65.81 - (0.1847 x heart rate (bpm)
Health-related quality of life | Baseline and 8-weeks
  Short Form 12 Health Survey (SF-12) Short Form 12 Health Survey (SF-12) Physical component score (PCS) 0-100 Mental component score (MCS) 0-100 The scores have a mean of 50 with a standard deviation of 10. Values above or below 50 indicate a better or worse state of physical or mental health.
Motivation to exercise | Baseline and 8-weeks
  Behavioural Regulation in Exercise Questionnaire-2 (BREQ-2). BREQ-2 has a Likert-type scale of 5 points, where 0 = not true for me and 4 = very true for me.
Exercise adherence | Baseline and 8-weeks
  Attendance at exercise sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No